CLINICAL TRIAL: NCT03332914
Title: A Crossover Designed Study to Evaluate Effects of Microcurrent Therapy on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Federal Ministry for Economic Affairs and Energy (Other)
Responsible Party: Principal Investigator, PD Dr. Martin Weigl, MPH, PD, MD, MPH (Harvard University), Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MicrocurrencyCrossover
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; microcurrent; knee; electrotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Active Comparator): control group fisrt and after washing out Microcurrent therapy: Channel A: 100µA; 200 Hz Duration of each treatment session: 30 minutes Number of sessions: 10
  Interventions: Device: Microcurrent therapy
- Second group (Active Comparator): Microcurrent therapy: Channel A: 100µA; 200 Hz Duration of each treatment session: 30 minutes Number of sessions: 10
  after washing out control group
  Interventions: Device: Microcurrent therapy

INTERVENTIONS:
Device: Microcurrent therapy — The microcurrent therapy will be applied with electrodes that are fixed around the knee. The two electrodes of channel A will be placed at the inner and outer side of the knee that is most affected by pain. The two electrodes of channel B will be placed above and below the patella. An apparatus with CE certificate will be used.

SUMMARY:
This crossover designed study evaluates the effects of microcurrent therapy on knee osteoarthritis. Ín a previous study patients were randomized into four different groups. Group 1 and 2 both received microcurrent therapy, but with different freqency and intensity parameters. Group 3 received treatment with the microcurrent treatment apparatus without current (sham). group 4 was a control group.

In the following, present study the controll group as well as the sham group will receive the microcurrent therapy (verum).

DETAILED DESCRIPTION:
The objective of the previous randomized, controlled pilot study was to evaluate the effect of microcurrent therapy on pain and physical function in patients with osteoarthritis of the knee. The secondary objective was to compare the effects of different currents. (group 1 - 4) After receiving 10 sessions of microcurrent therapy the statistical calculation showed a slightly significant difference in the verum-group A (Parameters Channel A: Channel B, Frequency ...) After a wash-out-phase we are now trying to evaluate and possibly confirm the positive effect of the previous trial. Therefore the control - and sham group from the previous study will now receive microcurrent therapy of apparatus A.

The whole procedure (Number of session, duration of the treatments, main outcome measurements, secondary outcome measurements) of the following study is identical with the previous pilot study. Assessments four the group will be at the first day of treatment (T1) and at the end of Treatment (T2).

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee
* pain intensity > 3 on the numerical rating scale (0-10)

Exclusion Criteria:

* knee arthroplasty
* gravity
* dermal Irritation at the skin of the knee
* carcinoma
* known osteoarthritis grade 4 (Kellgren and Lawrence score)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Numerical Rating scale (NRS) for pain (0-10) | Change of NRS: Before treatment vs. end of treatment (in average 21 days later)
  numerical Rating scale

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | Change of scores: Before treatment vs. end of treatment (in average 21 days later
  Knee specific Instrument measuring pan, function and Quality of life.
Short-Form 36 | Change of scores: Before treatment vs. end of treatment (in average 21 days later)
  Generic HRQOL measure
Satisfaction with Treatment (Questionnaire) | Evaluation at the end of treatment (in average 21 days after Start of treatment)
  Self-administered questionnaire that was developed for this study
Range of Motion knee joint | Change: Before treatment vs. end of treatment (in average 21 days later)
  Clinical test with goniometer
Get-up-and-Go-Test (GUG) | Change: Before treatment vs. end of treatment (in average 21 days later)
  clinical test that measures mobility
6-minute walking test | Change: Before treatment vs. end of treatment (in average 21 days later)
  Clinical test that measures the Walking ability

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwig Maximilian University, University Hosipital, Department of Orthopedics, Physical Medicine and Rehabilitation, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No